CLINICAL TRIAL: NCT02422446
Title: Effects of Eicosapentaenoic Acid on Endothelial Function in Diabetic Subjects: A Pilot Trial
Brief Title: Effects of Eicosapentaenoic Acid on Endothelial Function in Diabetic Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty enrolling patients with elevated triglycerides under statin treatment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Luc Djousse, Director of Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013D003968
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease
Keywords: Endothelial function; Eicosapentaenoic acid; Triglycerides
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — eicosapentaenoic acid ethyl ester; Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPA arm (Experimental): EPA arm will receive 4 grams per day of EPA (icosapent ethyl) taken twice a day
  Interventions: Drug: Icosapent ethyl
- Control (No Intervention): Control group will not receive EPA

INTERVENTIONS:
Drug: Icosapent ethyl — icosapent ethyl is eicosapentaenoic acid, an omega-3 fatty acid that naturally occurs in fish
  Other Names: Vascepa; Eicosapentaenoic Acid; EPA
  Arms: EPA arm

SUMMARY:
This pilot trial seeks to obtain preliminary data on the effects of eicosapentaenoic acid (EPA) (4g/d) on endothelial function measured via endopat2000 after 12 weeks of intervention among adults with elevated triglycerides and type 2 diabetes.

DETAILED DESCRIPTION:
Thirty adults aged 30-75 y will be randomized to either 4 g/d of eicosapentaenoic acid or no drug for 12 weeks. Endothelial function will be measured at baseline and after 12 weeks. in a secondary aims, we will evaluate effects of eicosapentaenoic acid (EPA) on plasma levels of c-reactive protein, oxidized low-density lipoprotein cholesterol, and endothelin-1.

ELIGIBILITY:
Inclusion Criteria:

* Age 30+ years
* Hypertriglyceridemia (150-400 mg/dl)
* Statin use for at least six months at the time of screening
* Type 2 diabetes treated with diet and/or oral hypoglycemic agents diagnosed 1+ year
* Ability to provide informed consent and provide blood samples
* Willingness to abstain from fish oil, EPA, over the counter niacin, and other omega-3 fatty acid supplements during the study period (12 weeks)
* Ability to travel to the study site at Brigham and Women's Hospital for 3 study visits
* Reactive hyperemia index (RHI) of ≤ 2.0

Exclusion Criteria:

* Eating disorder or heavy drinkers
* Treatment with chronic prescription pharmacotherapy for metabolic or cardiovascular disease management or risk factor modification
* Pregnant or lactating women
* Statin use <6 months at the time of screening
* Allergy to EPA, fish oil, or other omega-3 fatty acids
* Current use of insulin, cyclophosphamide, estrogen, fibrates, niacin, hormone replacement therapy, testosterone, oral contraceptives, growth hormones, insulin-like growth factor-1, and other systemic steroids.
* Inability to provide informed consent or blood samples
* History or prevalent diagnosis of cancer, asthma, kidney insufficiency, stroke, seizures, allergic disorders, or congestive heart failure
* Diagnosis of diabetes < 1 year prior to enrollment
* Intention to move out of greater Boston area within one year
* Current use of omega-3 supplements, fish oil, or >2 servings of fish per week
* Bleeding disorder or uncontrolled endocrine (i.e., thyroid) or metabolic disorders
* Treatment with blood thinning drugs (i.e. warfarin and clopidogrel)
* Major surgical operation 3 months before or after screening
* Organ transplantation
* Current participation in another trial or plan to do so during the study
* Inability to give informed consent or to travel to the study center at Brigham and Women's Hospital
* RHI of >2.0
* Triglycerides <150 mg/dl or >400 mg/dl
* Body mass index of 40+ kg/m2

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EPA Arm | Control
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EPA Arm | Control | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 69 [69 to 69] | 57 [57 to 57] | 63 [57 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Triglycerides [Mean (Full Range); unit: mg/dl] | 221 [221 to 221] | 177 [177 to 177] | 199 [177 to 221]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Endothelial Function at 12 Weeks Using Reactive Hyperemia Index (RHI)
Description: Digital pulse amplitude will be measured with a fingertip peripheral arterial tonometry (PAT) device (Endo-PAT2000, Itamar Medical) in a supine position. Baseline pulse amplitude will be measured for 5 minutes, then the arterial flow will then be interrupted for 5 minutes with a cuff placed on a proximal forearm. Pulse amplitude will be recorded electronically and analyzed by a computerized and automated algorithm. The change from the baseline measurement will be expressed as the reactive hyperemia index (RHI). We will calculate the pulse amplitude response to hyperemia for each 30-second interval as a ratio of the post-deflation pulse amplitude to the baseline pulse amplitude as described previously. The RHI ratio will be computed by dividing the ratio obtained on the test side over the ratio from the control finger. We will assess change in RHI ratio between baseline value and 12-week value after the intervention.
Time Frame: Between baseline and 12 weeks
Measure: Mean (Full Range); unit: % change from baseline value
Arm/Group | EPA Arm | Control
Number analyzed (Participants) | 1 | 1
% change from baseline value | -29 [-29 to -29] | -1.6 [-1.6 to -1.6]

2. Secondary Outcome: Change in Endothelin-1 (ET-1), High-sensitive C-reactive Protein (hsCRP), and Oxidized LDL Between Baseline and 12 Weeks
Description: Plasma hsCRP will be measured by Sandwich enzyme linked immunosorbent assay (ELISA). Plasma oxidized LDL and plasma ET-1 will be measured using a commercially available sandwich-enzyme immunoassay kit (R & D).
Time Frame: change between baseline and 12 weeks post-intervention
Population: Because the trial was terminated prematurely due to difficulties in finding suitable subjects, we were not able to measure any of the three biomarkers specified under the secondary outcome (ET-1, hsCRP, and Oxidized LDL).
Arm/Group | EPA Arm | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Total study period of 12 weeks
Arm/Group | EPA Arm | Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT02422446/Prot_SAP_002.pdf
  • Informed Consent Form (2015-05-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT02422446/ICF_003.pdf